CLINICAL TRIAL: NCT05767203
Title: Search for Genetic Markers and Biomarkers to Follow Patients With Intellectual Disabilities of Genetic Origin and to Understand Its Origin and Associated Comorbidities
Brief Title: Genetic Markers and Biomarkers in Patients With Intellectual Disabilities of Genetic Origin
Acronym: BioJeL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Jerome Lejeune (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BioJeL
Record Dates: First submitted 2023-02-07; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Down Syndrome; Intellectual Disability
MeSH Terms: conditions — Down Syndrome; Intellectual Disability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Down syndrome or other Intellectual deficiency of genetic origin (Experimental): Patients with Down syndrome or with other intellectual deficiency of genetic origin followed at the outpatients clinic of the Institut Jérôme Lejeune.
  Interventions: Other: Biological samplings

INTERVENTIONS:
Other: Biological samplings — Blood and/or skin samples

SUMMARY:
Analyze genetic and biological markers in patients with Intellectual Deficiencies (ID) of genetic origin in order to better understand the mechanisms of modified genes, cellular mechanisms, pathways involved in different disorders , complications and pathologies associated with ID of genetic origin.

DETAILED DESCRIPTION:
Blood and skin samples will be taken from patients coming at the outpatients clinic of the Institut Jérôme Lejeune and who consent to participate to the study. Search and identification of markers will be then done from the collected samples.

ELIGIBILITY:
Inclusion Criteria:

* Patient diagnosed with an intellectual disability of genetic origin
* Patient of all ages coming for consultation at the Institut Jérôme Lejeune
* Patient whose parents or legal representative have received and understood the information document and signed the informed consent for a sample for the research project.
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Parents unable to find out about the constraints related to the study
* Refusal of informed patient participation
* Pregnant, parturient and nursing mothers
* Persons deprived of their liberty by judicial or administrative decision

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2032-09-01 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of biomarkers in blood | 10 years
  Analysis of biomarkers from blood samples taken during the visit
Identification of biomarkers from skin samples | 10 years
  Analysis of biomarkers from skin samples taken during the visit

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Jérôme Lejeune, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided